CLINICAL TRIAL: NCT04241978
Title: The Effectiveness of a Web-based Decision Aid for Patients With Hip Osteoarthritis: Study Protocol for a Randomized Controlled Trial
Brief Title: Development and Evaluation of a Web Based Decision Aid for Patients With Hip Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Servicio Canario de Salud (Other)
Collaborators: Fundación Canaria de Investigación Sanitaria (Other); Hospital Universitario de Canarias (Other); Hospital San Juan de Dios Tenerife (Other); Avedis Donabedian Research Institute (Other); Gerencia de Atención Primaria del Área de Salud de Tenerife (Unknown)
Responsible Party: Principal Investigator, Lilisbeth Perestelo-Perez, Health Services Researcher, Servicio Canario de Salud
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PIFUN33/18
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Hip Osteoarthritis; Osteoarthritis
Keywords: Hip osteoarthritis; Patient decision aids; Person-centred care; Randomized controlled trial; Shared decision-making; Web-based intervention
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The participants will complete the baseline assessment and will be asked to read the project information sheet. Then, patients allocated to the intervention group will review the PtDA accompanied by the researcher and will complete the questionnaires assessing the outcome measures, in the same web interface.
  Interventions: Other: Patient Decision Aid (PtDA)
- Control group (Active Comparator): Patients in the control group will follow the same procedure, but they will be given a brochure with general information about osteoarthritis of the hip, knee, ankle and foot instead of the PtDA
  Interventions: Other: Brochure with general information about osteoarthritis

INTERVENTIONS:
Other: Patient Decision Aid (PtDA) — Patient Decision Aid (PtDA) are tools that enables to promote and facilitate patients' involvement in medical decisions concerning their health
  Other Names: Intervention
  Arms: Intervention group
Other: Brochure with general information about osteoarthritis — Participants of the control group will be given a brochure with general information about osteoarthritis of the hip, knee, ankle and foot instead of the PtDA
  Other Names: Control
  Arms: Control group

SUMMARY:
The main goal of this study is assess the effectiveness of a PtDA for patients with hip osteoarthritis

DETAILED DESCRIPTION:
Background: Osteoarthritis (OA) is a health condition sensitive to patient's preferences and values regarding the benefits and risks of the different treatment options. In this sense, patient decision aids (PtDA) can play an important role in helping patients to incorporate their values, needs and preferences into the decision-making process, thus improving Person-Centred Care (PCC). Previous research has focused almost exclusively on knee OA, and therefore the aim of this study is to develop and evaluate the effectiveness of a PtDA for patients with hip OA.

Methods: The general design consists of two phases: 1) design a web-based PtDA for patients with hip OA, following the recommended procedures: systematic review of safety/effectiveness of treatments, and an iterative process of development with the help of an Advisory Committee composed of health professionals and patients; 2) To evaluate the impact of the PtDA on hip OA patients' decision-making process related with their treatment. For that aim, a multicenter randomized controlled trial will be carried out with 124 patients with hip OA in Tenerife (Spain) comparing intervention or usual care.

Discussion: PtDAs have been recommended as a useful and effective resource for improving PCC in many health conditions. The intervention is intended to empower patients by fostering their active participation during the decision-making process about their treatment, and by ensuring they make informed decisions congruent with their values and preferences. This study will contribute to the scientific knowledge about effectiveness of PtDAs in hip OA, in order to improve the quality of health care offered to these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of hip Osteoarthritis

Exclusion Criteria:

* Patients younger than 18 years
* Previous hip arthroplasty
* Patients with terminal illnesses
* Non-fluent Spanish language
* Mental or sensory alterations that impede or hinder the response to the measurement instruments or do not have the capacity to make decisions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Decisional conflict regarding the treatment for Hip Osteoarthritis, measured by the Decisional Conflict Scale (DCS) | Immediately after the intervention
  DCS is a 16-item self-reported scale widely used in PtDA research. It is composed of five subscales: uninformed, values, support, uncertainty and effectiveness. This is a 0-100 point scale, where a high score means more decisional conflict.

SECONDARY OUTCOMES:
Knowledge of the disease and treatments | Before and immediately after the intervention
  A 7-item scale will be udes to assess patients' knowledge of the disease and treatments
Values about characteristics of treatments | Immediately after the intervention
  Patients will be asked to rate in a 0-10 scale the importance they attribute to different characteristics of treatment: mode of administration, improvement in pain and function, risk of mild and serious adverse effects, time until symptoms' improvement, duration of benefits, and in the case of arthroplasty, period of rehabilitation and risk of needing surgery revision.
Treatment preference | Immediately after the intervention
  Patients will be asked the treatment they prefer: physiotherapy, medication, intra-articular injections, arthroplasty, not sure
Intention to undergo the preferred treatment | Immediately after the intervention
  Assessed with one item ranging 0 (not sure) to 5 (completely sure)
Concordance between values and intention to undergo arthroplasty vs. conservative treatments | Immediately after the intervention
  Binary variable (yes/no) derived from the association between values and intention to undergo arthroplasty (see statistical analysis).
Decision quality about arthroplasty | Immediately after the intervention
  Binary variable (yes/no) defined as a combination of adequate knowledge (≥60% of correct responses) and concordance.
Satisfaction with the decision making process scale | Immediately after the intervention
  The Satisfaction with Decision Scale (SWD) is a validated 12-item scale measuring participants' satisfaction with healthcare decision making. The SWD uses a 5-point Likert scale where 0 is "Strongly Disagree" and 4 is "Strongly Agree." This is a 0-100 point scale, where a high score means more satisfaction with the decision making process.

CONTACTS AND LOCATIONS:
Overall Officials: Lilisbeth Perestelo Perez, PhD, Principal Investigator — Servicio de Evaluación de. Servicio Canario de Salud
Locations (1):
- Evaluation Unit. Canary Islands Health Service, Santa Cruz de Tenerife, Santa Cruz Tenerife, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perestelo-Perez L, Alvarez-Perez Y, Rivero-Santana A, Ramos-Garcia V, Duarte-Diaz A, Torres-Castano A, Toledo-Chavarri A, Herrera-Perez M, Pais-Brito JL, Del Castillo JC, Vazquez JR, Orrego C, Serrano-Aguilar P. The effectiveness of a web-based decision aid for patients with hip osteoarthritis: study protocol for a randomized controlled trial. Trials. 2020 Aug 24;21(1):736. doi: 10.1186/s13063-020-04661-z. PMID 32838800